## **FENUGREEK: AN EMERGENT ALLERGEN**

NCT ID not yet assigned

**DATE: January 15, 2024** 



University hospital Polyclinic "G. Martino" - Messina

## **OPERATIVE UNIT OF ALLERGY AND CLINICAL IMMUNOLOGY**

## INFORMED CONSENT FOR THE PROCESSING OF CLINICAL DATA FOR RESEARCH USE

| I, the undersigned(patient first and last name) |
|---|
| bornresident in, |
| DECLARE TO |
| have been informed that all personal and clinical data collected, will be considered |
| have been informed that all personal and clinical data collected, will be considered confidential and stored in compliance with applicable privacy laws. |
| communication and society in compilation with applicable privacy laws. |
| I also: • AGREE • DO NOT AGREE |
| to the utilization of clinical data, including photographic or filmed images, related to the |
| health care services being processed in an anonymous form for research, epidemiology, |
| education, and disease study aims. |
| Messina, (date) |
| Patient signature |
| Tuttent signature |